CLINICAL TRIAL: NCT05848466
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BAT8010 for Injection in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Assessment of Safety, Tolerability and Pharmacokinetics With BAT8010 for Injection in Advanced Malignant Solid Tumors Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8010-001-CR
Record Dates: First submitted 2023-02-06; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-02

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A/ Accelerated titration 0.8mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 0.8mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- B/ Standard 3+3 1.2mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 1.2mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- C/ Standard 3+3 2.4mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 2.4mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- D/ Standard 3+3 3.6mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 3.6mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- E/ Standard 3+3 4.8mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 4.8mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- F/ Standard 3+3 6.0mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 6.0mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- G/ Standard 3+3 7.2mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 7.2mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection
- H/ Standard 3+3 8.4mg/kg of BAT8010 (Experimental): Drug: BAT8010, Dosage: 8.4mg/kg, Frequency: once every 3 weeks, Duration: 1year
  Interventions: Drug: BAT8010 for Injection

INTERVENTIONS:
Drug: BAT8010 for Injection — Intravenous

SUMMARY:
The goal of this interventional study is to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of BAT8010 for injection in patients with advanced or metastatic solid tumors, explore the maximum tolerable dose. Participants will be given one of below dose once every three weeks: 0.8mg/kg, 1.2mg/kg, 2.4mg/kg, 3.6mg/kg, 4.8mg/kg, 6.0mg/kg, 7.2mg/kg, 8.4mg/kg. The dose escalation follow adopt accelerated titration and "3+3" dose increasing rule.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent.
* The expected survival period is more than 3 months base on the evaluation of the investigator.
* Eastern Cooperative Oncology Group (ECOG) should be 0-1.
* Patients who fail to standard treatment or have no standard treatment or are not suitable for standard treatment at this stage, and who have Human epidermal growth factor receptor-2 (HER2) expression (including Immunohistochemistry (IHC)3+, IHC2+/fluorescence in situ hybridization (FISH)+and IHC2+/FISH - patients) confirmed by histopathology and cytopathology, the dose escalation stage includes but is not limited to breast cancer, gastric cancer, non-small cell lung cancer, biliary tract cancer, colorectal cancer, urothelial cancer, etc., and the expansion stage only includes breast cancer.
* An evaluable tumor focus was necessary in the dose escalation stage, and at least one measurable tumor focus in the dose expanding stage (according to RECIST 1.1 standard).
* Enough organs, bone marrow reserve function and heart function.
* Must agree to take effective contraceptive methods to prevent pregnancy.

Exclusion Criteria:

* Previously received HER2 targeted drug therapy such as trastuzumab or pertuzumab, Trastuzumab Emtansine or Enhertu, and the treatment of topoisomerase I inhibitors (such as irinotecan), there were adverse event (AE) equal to or pass 3 levels that were determined to be treatment-related or drug related
* Before the first administration of the investigational drug, the AE (CTCAE5.0) caused by previous anti-tumor treatment was still higher than grade 1
* Primary central nervous system tumor or symptomatic central nervous system metastasis, meningeal metastasis or previous history of epilepsy. Patients with asymptomatic or symptomatic central nervous system metastasis who have achieved clinical control but are judged stable by the investigator can be included.
* Major surgery has been performed within 28 days before the first use of the study drug, or if it has been more than 21 days after surgery, but the postoperative complications are still continuing.
* Subjects who had severe infection within 4 weeks before the first administration, or had any symptoms and signs of active infection within 2 weeks before the first administration.
* Untreated or under treatment tuberculosis subjects, with a history of immune deficiency, or other immune deficiency diseases, or with a history of organ transplantation.
* Active hepatitis B virus infected, hepatitis C virus infected, Treponema pallidum antibody positive and Rapid plasma reagin ring card test (RPR) positive.
* Patients with symptomatic congestive heart failure (New York Heart Association (NYHA) grade II to IV) or serious arrhythmia requiring treatment (QTc prolongation of 12-lead electrocardiogram (ECG) 450 ms [male], 470 ms [female]), and patients with myocardial infarction and unstable angina pectoris in the past 6 months. Except for atrial fibrillation or paroxysmal supraventricular tachycardia
* Patients who have a history of non-infectious pneumonia requiring glucocorticoid treatment or who currently have interstitial lung disease.
* There are any other serious potential diseases.
* Previous anti-tumor therapy (such as chemotherapy, endocrine therapy, targeted therapy, immunotherapy or tumor embolization) is less than 28 days from the first study administration.
* Therapeutic radiopharmaceuticals must be discontinued 8 weeks before the first study administration.
* Known allergy or intolerance to the study drug or its excipients.
* Pregnant or lactating women.
* The study participants who were considered unsuitable for the study by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 3 weeks
  Grade 5 toxicity; Hematological toxicity: Grade 4 alanine-aminotransferase(ALT) or aspartate-aminotransferase(AST) increase: AST or ALT>5 times upper limit of normal value(ULN), with ≥ 2 levels of blood bilirubin increase; Hematological toxicity: Grade 4 neutropenia lasting>7 days. ≥Grade 3 neutropenia with fever (single body temperature>38.3 or continuous body temperature ≥ 38 ℃, more than 1 Hour). Grade 4 anemia. Grade 4 thrombocytopenia. ≥ Grade 3 thrombocytopenia and lasting>7 days. ≥ Grade 3 thrombocytopenia with bleeding; Other ≥Grade 3 non hepatic toxicity, non hematological toxicity.
maximum tolerated dose (MTD) | 3 weeks
  MTD was defined as the highest dose level of DLT observed in ≤1/6 subjects in a dose group during the DLT evaluation period

SECONDARY OUTCOMES:
Pharmacokinetic | every cycle until 18 weeks (one cycle equals 3 weeks)]
  Cmax
Immunogenicity | every cycle until 18 weeks, every 4 cycles after 18 weeks (one cycle equals 3 weeks), up to 1 year
  Presence of anti drug antibody (ADA)/Neutralizing antibodies (NAb) ADA, Nab
Objective response rate (ORR) | through study completion, an average of 2 years
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and remained for a certain period of time, including CR and PR cases. Specifically divided into: 1.The ratio of patients with partial response (PR) or complete remission (CR) efficacy at the end of the first 6 cycles (18 weeks) of treatment. 2.The proportion of patients whose best response reached PR or CR during the entire study period.
Duration of remission (DoR) | Through study completion, an average of 2 years
  DoR is defined as the time between the first assessment of objective remission of a tumor and death from any cause before the first assessment of Disease progression (PD) , reflecting the duration of ORR.
Disease Control Rate (DCR) | through study completion, an average of 2 years
  The proportion of patients with reduced or stable tumors that remain for a certain period of time, including CR, PR, and Disease stability (SD) cases.
Progression free survival (PFS) | through study completion, an average of 2 years
  The time from the first administration to the occurrence of objective tumor progression or all cause death
Total survival period (OS) | through study completion, an average of 2 years
  The time from the date of first administration to the occurrence of death due to any cause. Subjects who were still alive at the time of analysis will use the date of their last contact as the deadline.

CONTACTS AND LOCATIONS:
Overall Officials: Chaohe Wang, Study Director — Bio-Thera Solutions
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No